CLINICAL TRIAL: NCT00142324
Title: A Randomised Placebo Controlled Trial of a Cholinesterase Inhibitor in the Management of Agitation in Dementia That is Unresponsive to a Psychological Intervention
Brief Title: CALM-AD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institute of Psychiatry, London (Other)
Collaborators: Medical Research Council (Other Government); Alzheimer's Society (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: ISRCTN62185868
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2005-12-14 (Estimated); Status verified 2005-09

CONDITIONS: Alzheimer's Disease
Keywords: Dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — Donepezil

INTERVENTIONS:
Drug: Donepezil

SUMMARY:
Primary Aim

To determine whether;

* Donepezil is significantly better than placebo in the management of agitation in Alzheimer's Disease that has not responded to, or is inappropriate for a standardised brief psychosocial treatment

Secondary Aims

To determine whether;

* Donepezil has a significant positive or negative impact upon quality of life compared with placebo
* whether there is a significant difference between Donepezil and placebo with respect to cognitive performance
* the cost effectiveness of the pharmacological treatment for agitation

ELIGIBILITY:
Inclusion Criteria: a diagnosis of dementia consistent with Diagnostic and Statistical Manual of Mental Health Disorders, revised 3rd edition (DSM-III-R) (APA, 1987) National Institute of Neurological and Communicative Disorders and Stroke - Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) diagnostic criteria for probably or possible AD (MKhann et al, 1984) (Appendix 6) clinically significant agitation (defined as causing distress to patient and at least moderate management problems for carers on at least two days per week for a two week period, together with a Cohen Mansfield Agitation Inventory (CMAI) (Cohen-Mansfield, 1986) (Appendix 11 A) score >39 age >39 years resident in care facility or community living with a carer not receiving treatment with neuroleptics or cholinesterase inhibitors currently or in the past four weeks and responsible clinician not considering treatment with cholinesterase inhibitor for the next 16 weeks taking into account the clinical evidence base and NICE guideline (NICE, 2001) patient with capacity willing to consent to study or will to participate in study if lacking capacity carer with capacity willing to consent to study and in agreement for patient lacking capacity to participate if patient willing to participate

-

Exclusion Criteria:known sensitivity to Donepezil severe, unstable or uncontrolled medical conditions apparent from history, physical examination or investigations current evidence of delirium patient meets criteria for Probably Dementia with Lewy Bodies (McKeith et al, 1996) low probability of treatment compliance

-

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 190
Dates: Start 2003-11; Study Completion 2005-12

PRIMARY OUTCOMES:
Cohen Mansfield Agitation Inventory

SECONDARY OUTCOMES:
Neuropsychiatric Inventory
Standardized Mini-Mental State Examination
Severe Impairment Battery
Clinical Global Impression of Severity/Change

CONTACTS AND LOCATIONS:
Overall Officials: Robert Howard, Principal Investigator — Institute of Psychiatry, London; Peter Bentham, Principal Investigator — Queen Elizabeth Psychiatric Hospital, Birmingham; Richard Brown, Principal Investigator — Institute of Psychiatry, London; Roger Bullock, Principal Investigator — Kingshill Research Centre, Victoria Hospital, Swindon; Alistair Burns, Principal Investigator — Wythenshawe Hospital, Manchester; Clive Holmes, Principal Investigator — Moorgreen Hospital, Southampton; Robin Jacoby, Principal Investigator — Warneford Hospital, Oxford; James Lindesay, Principal Investigator — Leicester General Hospital, Leicester; John O'Brien, Principal Investigator — Newcastle General Hospital, Newcastle
Locations (8):
- United Kingdom (8):
  - Queen Elizabeth Psychiatric Hospital, Birmingham
  - Department of Psychiatry for the Elderly, Leicester General Hospital, Leicester
  - Institute of Psychiatry, King's College, London, London
  - Old Age Psychiatry, Wythenshawe Hospital, Manchester, Manchester
  - Institute for Ageing and Health, Newcastle General Hospital, Newcastle, Newcastle upon Tyne
  - Department of Psychiatry, Warneford Hospital, Oxford, Oxford
  - MARC, Moorgreen Hospital, Southamptom, Southampton
  - Department of Old Age Psychiatry, Victoria Hospital, Swindon, Swindon

REFERENCES:
- [Derived] Howard RJ, Juszczak E, Ballard CG, Bentham P, Brown RG, Bullock R, Burns AS, Holmes C, Jacoby R, Johnson T, Knapp M, Lindesay J, O'Brien JT, Wilcock G, Katona C, Jones RW, DeCesare J, Rodger M; CALM-AD Trial Group. Donepezil for the treatment of agitation in Alzheimer's disease. N Engl J Med. 2007 Oct 4;357(14):1382-92. doi: 10.1056/NEJMoa066583. PMID 17914039